CLINICAL TRIAL: NCT00104858
Title: Nonmyeloablative Conditioning With Pre- and Post-Transplant Rituximab Followed by Related or Unrelated Donor Hematopoietic Cell Transplantation for Patients With Advanced Chronic Lymphocytic Leukemia: A Multi-Center Trial
Brief Title: Fludarabine Phosphate, Radiation Therapy, and Rituximab in Treating Patients Who Are Undergoing Donor Stem Cell Transplant Followed by Rituximab for High-Risk Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1840.00; NCI-2009-01594 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1840.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA018029 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-06

CONDITIONS: Chronic Lymphocytic Leukemia; Prolymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Stage III Chronic Lymphocytic Leukemia; Stage III Small Lymphocytic Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Small Lymphocytic Lymphoma; T-Cell Large Granular Lymphocyte Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic; Leukemia, Large Granular Lymphocytic | interventions — Cyclosporine; Cyclosporins; fludarabine phosphate; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Rituximab; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Patients receive a conditioning regimen comprising fludarabine IV on days -4 to -2 and rituximab IV on days -3, 10, 24, and 38.
  Patients undergo single fraction low-dose TBI on day 0. After completion of TBI, patients undergo allogeneic hematopoietic stem cell transplantation on day 0. Patients then receive rituximab IV on days 10, 24, and 38.
  Patients receive an immunosuppressive regimen comprising cyclosporine PO BID on days -3 to 56 followed by a taper to day 180 (related recipients) or on days -3 to 100 followed by a taper to day 180 (unrelated recipients). Patients also receive mycophenolate mofetil PO BID on days 0-27 (related recipients) or TID on days 0-40 followed by a taper to day 96 (unrelated recipients).
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclosporine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Pharmacological Study; Biological: Rituximab; Radiation: Total-Body Irradiation

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo HSCT
  Other Names: allogeneic stem cell transplantation; HSC; HSCT
Drug: Cyclosporine — Given PO
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Gengraf; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; Oforta; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo HSCT
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation
Other: Pharmacological Study — Correlative studies
Biological: Rituximab — Given IV
  Other Names: BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar BI 695500; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; RTXM83
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation

SUMMARY:
This phase II trial studies how well fludarabine phosphate with radiation therapy and rituximab followed by donor stem cell infusions work in treating patients with high-risk chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) with low side effects. Nonmyeloablative stem cell transplants use low doses of chemotherapy (fludarabine phosphate) and radiation to suppress the patient's immune system enough to prevent rejection of the donor's stem cells. Following infusion of donor stem cells, a mixture of the patient's and the donor's stem cells will exist and is called "mixed chimerism". Donor cells will attack the patient's leukemia. This is called the "graft-versus-leukemia" effect. Rituximab will be given 3 days before and three times after infusing stem cells to help in controlling CLL early after transplant till the "graft-versus-leukemia" takes control. Further, rituximab could augment the "graft-versus-leukemia" effect by activating donor immune cells and hence improve disease control. Sometimes the transplanted cells from a donor can also attack the body's normal cells. Giving cyclosporine and mycophenolate mofetil after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether nonmyeloablative conditioning and allogeneic hematopoietic cell transplantation (HCT) improves survival at 18 months for patients with fludarabine (fludarabine phosphate)-refractory, fludarabine/cyclophosphamide/rituximab (FCR)-failed, or del 17p CLL over that of historical controls (45% at 18 months) given CAMPATH-1H (alemtuzumab).

SECONDARY OBJECTIVES:

I. Estimate the overall response rate (complete remission [CR] + partial remission [PR]) by standard morphologic, flow cytometric, and molecular techniques.

II. Assess the rate of relapse/progression.

III. Define incidences of regimen-related toxicities (RRT) and infections within the first 100 days and the incidence of transplant-related mortality (TRM) within the first year.

IV. Estimate incidences of grade II-III and III-IV acute graft-versus-host disease (GVHD) and chronic GVHD.

V. Determine whether the addition of rituximab to the nonmyeloablative conditioning and allogeneic HCT improves survival at 18 months over our historical data (57% at 18 months).

VI. Determine the incidence of serious adverse events with the addition of rituximab in comparison to historical data of unrelated nonmyeloablative HCT.

VII. Evaluate the pharmacokinetics of rituximab.

VIII. Evaluate B-cell and T-cell immune reconstitution in comparison to historical data of unrelated nonmyeloablative HCT.

IX. Describe donor and host polymorphisms of the FCgammaRIIIa receptor and cluster of differentiation (CD)32 and evaluate their impact on disease response and relapse.

X. Investigate the mechanism of disease resistance in relapsed/nonresponding patients.

XI. Isolate donor cytotoxic T lymphocytes specific for host minor histocompatibility antigens.

OUTLINE:

Patients receive a conditioning regimen comprising fludarabine phosphate intravenously (IV) on days -4 to -2 and rituximab IV on days -3, 10, 24, and 38.

Patients undergo single fraction low-dose total-body irradiation (TBI) on day 0. After completion of TBI, patients undergo allogeneic hematopoietic stem cell transplantation (HSCT) on day 0. Patients then receive rituximab IV on days 10, 24, and 38.

Patients receive an immunosuppressive regimen comprising cyclosporine orally (PO) twice daily (BID) on days -3 to 56 followed by a taper to day 180 (related recipients) or on days -3 to 100 followed by a taper to day 180 (unrelated recipients). Patients also receive mycophenolate mofetil PO BID on days 0-27 (related recipients) or three times daily (TID) on days 0-40 followed by a taper to day 96 (unrelated recipients).

After completion of study treatment, patients are followed up at 6 months, 1 year, 18 months, 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of CLL (or SLL) or diagnosis of CLL that progresses to prolymphocytic leukemia (PLL)
* Patients with B-Cell CLL or PLL who:

  * Failed to meet National Cancer Institute (NCI) Working Group criteria 2 for complete or partial response after 2 cycles of therapy with regimen containing fludarabine (or another nucleoside analog, e.g. cladribine [2-CDA], pentostatin) or with disease relapse within 12 months after completing therapy with a fludarabine (or another nucleoside analog) containing regimen
  * Failed FCR or pentostatin/cyclophosphamide/rituximab (PCR) combination chemotherapy at any time point
  * Patients with novo or acquired "17p deletion" cytogenetic abnormality; patients should have received induction treatment but could be transplanted in 1st CR
* Patients who have suitable human leukocyte antigen (HLA)-matched related or unrelated donors willing to receive filgrastim (G-CSF), undergo leukapheresis to collect peripheral blood mononuclear cell (PBMC), and to donate stem cells
* RELATED DONORS: When more than one potential donor exists, priority should be given to donors based on HLA identity > cytomegalovirus (CMV) seronegativity > ABO compatibility > sex matching

  * Donor who is HLA phenotypically or genotypically identical at the allele level at HLA-A, -B, -C, -DRB1, and -DQB1
  * Must consent to G-CSF administration and leukapheresis;
  * Must have adequate veins for leukapheresis or agree to placement of central venous catheter (femoral, subclavian);
  * Only G-CSF mobilized PBMC only will be permitted as a hematopoietic stem cell (HSC) source on this protocol
* UNRELATED DONORS:

  * Fred Hutchinson Cancer Research Center (FHCRC) matching allowed will be Grades 1.0 to 2.1; Unrelated donors who are prospectively:
  * Matched for HLA-A, B, C, DRB1 and DQB1 by high resolution typing
  * Only a single allele disparity will be allowed for HLA-A, B, or C as defined by high resolution typing
* UNRELATED DONORS: Donors are excluded when preexisting immunoreactivity is identified that would jeopardize donor hematopoietic cell engraftment; this determination is based on the standard practice of the individual institution; recommended procedure for patients with 10 of 10 HLA allele level (phenotypic) match is to obtain a panel reactive antibody screens to class I and II antigens for all patients before HCT; if the PRA shows > 10% activity, then flow cytometric or B and T cell cytotoxic cross matches should be obtained; the donor should be excluded if any of the cytotoxic cross match assays are positive; for those patients with an HLA Class I allele mismatch, flow cytometric or B and T cell cytotoxic cross matches should be obtained regardless of the PRA results; a positive anti-donor cytotoxic crossmatch is an absolute donor exclusion
* UNRELATED DONORS: Patient and donor pairs homozygous at a mismatched allele in the graft rejection vector are considered a two-allele mismatch, i.e., the patient is A*0101 and the donor is A*0102, and this type of mismatch is not allowed
* UNRELATED DONORS: Only G-CSF mobilized PBMC will be permitted as a HSC source on this protocol

Exclusion Criteria:

* Infection with human immunodeficiency virus (HIV)
* Active diagnosis of central nervous system (CNS) involvement with CLL
* Patients unwilling to use contraceptive techniques before and for 12 months after HCT
* Pregnant women or females who are breastfeeding
* The addition of cytotoxic agents for 'cytoreduction' with the exception of tyrosine kinase inhibitors (such as imatinib mesylate), cytokine therapy, hydroxyurea, low dose cytarabine, chlorambucil, or rituxan will not be allowed within three weeks of the initiation of conditioning
* Active bacterial or fungal infections unresponsive to medical therapy
* Performance status: Karnofsky score < 60 for adult patients
* Cardiac ejection fraction < 40%; ejection fraction is required if age > 50 years or there is a history of prior transplant, anthracycline exposure or history of cardiac disease; and poorly controlled hypertension despite multiple antihypertensives
* Diffusing capacity of the lung for carbon monoxide (DLCO) < 40%, total lung capacity (TLC) < 40%, forced expiratory volume in 1 second (FEV1) < 40% and/or requiring continuous supplementary oxygen, or severe deficits in pulmonary function testing as defined by pulmonary consultant service; and the FHCRC principal investigator (PI) of the study must approve of enrollment of all patients with pulmonary nodules
* Patients with clinical or laboratory evidence of liver disease would be evaluated for the cause of liver disease, its clinical severity in terms of liver function, and the degree of portal hypertension; patients will be excluded if they are found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, hepatic damage with bridging fibrosis, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices or hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dl, or symptomatic biliary disease
* Patients with active non-hematologic malignancies (except non-melanoma skin cancers); this exclusion does not apply to patients with non-hematologic malignancies that do not require therapy
* Patients with a history of non-hematologic malignancies (except non-melanoma skin cancers) currently in a complete remission, who are less than 5 years from the time of complete remission, and have a > 20% risk of disease recurrence; this exclusion does not apply to patients with non-hematologic malignancies that do not require therapy
* DONOR: Age < 12 years
* DONOR: Identical twin
* DONOR: Pregnancy
* DONOR: Infection with HIV
* DONOR: Inability to achieve adequate venous access
* DONOR: Known allergy to filgrastim (G-CSF)
* DONOR: Current serious systemic illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2004-12 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Sorror, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (5):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - VA Puget Sound Health Care System, Seattle, Washington
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
- Rigshospitalet University Hospital, Copenhagen, Denmark
- University of Torino, Torino, Italy

REFERENCES:
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Chemotherapy and Rituximab Followed by HCT): Patients receive a conditioning regimen comprising fludarabine IV on days -4 to -2 and rituximab IV on days -3, 10, 24, and 38.
  Patients undergo single fraction low-dose TBI on day 0. After completion of TBI, patients undergo allogeneic hematopoietic stem cell transplantation on day 0. Patients then receive rituximab IV on days 10, 24, and 38.
  Patients receive an immunosuppressive regimen comprising cyclosporine PO BID on days -3 to 56 followed by a taper to day 180 (related recipients) or on days -3 to 100 followed by a taper to day 180 (unrelated recipients). Patients also receive mycophenolate mofetil PO BID on days 0-27 (related recipients) or TID on days 0-40 followed by a taper to day 96 (unrelated recipients).
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo HSCT
  Cyclosporine: Given PO
  Fludarabine Phosphate: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given PO
  Peripheral Blood Stem Cell Transplantation:
Period: Overall Study
Arm/Group | Treatment (Chemotherapy and Rituximab Followed by HCT)
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Historical Controls were utilized for comparison
Groups:
- Treatment: Patients receive fludarabine intravenously (IV) on days -4 to -2 and rituximab IV on days -3, 10, 24, and 38.
  Patients undergo single fraction low-dose total-body irradiation (TBI) on day 0. After completion of TBI, patients undergo allogeneic hematopoietic stem cell transplantation (HSCT) on day 0.
  Patients receive an immunosuppressive regimen comprising cyclosporine orally (PO) twice daily (BID) on days -3 to 56 followed by a taper to day 180 (related recipients) or on days -3 to 100 followed by a taper to day 180 (unrelated recipients). Patients also receive mycophenolate mofetil PO BID on days 0-27 (related recipients) or three times daily (TID) on days 0-40 followed by a taper to day 96 (unrelated recipients).
Arm/Group | Treatment
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 11
Age, Continuous [Median (Full Range); unit: years] | 59.5 [35 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 51
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 41
  Denmark | 7
  Italy | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Number of participants surviving post-transplant
Time Frame: At 18 months
Population: 14 subjects were enrolled prior to the addition of rituximab. These subjects are counted towards accrual but not evaluated with respect to outcome measures.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Chemotherapy and Rituximab Followed by HCT): Patients receive a conditioning regimen comprising fludarabine IV on days -4 to -2 and rituximab IV on days -3, 10, 24, and 38.
  Patients undergo single fraction low-dose TBI on day 0. After completion of TBI, patients undergo allogeneic hematopoietic stem cell transplantation on day 0. Patients then receive rituximab IV on days 10, 24, and 38.
  Patients receive an immunosuppressive regimen comprising cyclosporine PO BID on days -3 to 56 followed by a taper to day 180 (related recipients) or on days -3 to 100 followed by a taper to day 180 (unrelated recipients). Patients also receive mycophenolate mofetil PO BID on days 0-27 (related recipients) or TID on days 0-40 followed by a taper to day 96 (unrelated recipients).
Arm/Group | Treatment (Chemotherapy and Rituximab Followed by HCT)
Number analyzed (Participants) | 52
Participants | 34

2. Secondary Outcome: Comparison of Survival, Serious Adverse Events, and B-cell and T-cell Immune Reconstitution With Historical Data
Time Frame: At 18 months
Population: Lack of funds to support sample collection analysis
Groups:
- Treatment (Chemotherapy Followed by HCT): Patients receive a conditioning regimen comprising fludarabine IV on days -4 to -2.
  Patients undergo single fraction low-dose TBI on day 0. After completion of TBI, patients undergo allogeneic hematopoietic stem cell transplantation on day 0.
  Patients receive an immunosuppressive regimen comprising cyclosporine PO BID on days -3 to 100 followed by a taper to day 180. Patients also receive mycophenolate mofetil PO TID on days 0-40 followed by a taper to day 96.
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo HSCT
  Cyclosporine: Given PO
  Fludarabine Phosphate: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given PO
  Peripheral Blood Stem Cell Transplantation:
Arm/Group | Treatment (Chemotherapy and Rituximab Followed by HCT) | Treatment (Chemotherapy Followed by HCT)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With Relapse/Progression
Description: Relapse/Progression criteria for CLL
  Progressive disease:
  ≥1 of: Physical exam/imaging studies ≥50% increase or new, circulating lymphocytes by morphology and/or flow cytometry ≥50% increase, and lymph node biopsy w/ Richter's transformation.
  Relapsed disease:
  Criteria of progression occurring 6 months after achievement of complete or partial remission.
Time Frame: Day 84
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy and Rituximab Followed by HCT)
Number analyzed (Participants) | 52
Participants | 1

4. Secondary Outcome: Graft-versus-leukemia Analysis by Mechanism of Disease Resistance in Relapsed or Non-responding Patients and Isolation of Donor Cytotoxic T Lymphocytes Specific for Host Minor Histocompatibility Antigens
Time Frame: Day 84
Population: Lack of funds to support sample collection and analysis
Arm/Group | Treatment (Chemotherapy and Rituximab Followed by HCT) | Treatment (Chemotherapy Followed by HCT)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Grade II-III and III-IV Acute GVHD and Chronic GVHD
Description: Number of patients who developed acute GVHD post-transplant. Grade I +1 to +2 skin rash, No gut or liver involvement Grade II +1 to +3 skin rash, +1 gastrointestinal involvement and/or +1 liver involvement Grade III +2 to +4 gastrointestinal involvement and/or +2 to +4 liver involvement with or without a rash Grade IV Pattern and severity of GVHD similar to grade 3 with extreme constitutional symptoms or death
  The diagnosis of chronic GVHD requires at least one manifestation that is distinctive for chronic GVHD as opposed to acute GVHD. In all cases, infection and others causes must be ruled out in the differential diagnosis of chronic GVHD.
Time Frame: Up to 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy and Rituximab Followed by HCT)
Number analyzed (Participants) | 52
Participants | 46

6. Secondary Outcome: Number of Participants With Regimen-related Toxicity and Infections
Description: Reported using the adapted National Cancer Institute Common Toxicity Criteria.
Time Frame: Within the first 100 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy and Rituximab Followed by HCT)
Number analyzed (Participants) | 52
Participants | 48

7. Secondary Outcome: Number of Participants With Treatment-related Mortality
Description: Number of subjects expired without disease progression/relapse.
Time Frame: Up to 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy and Rituximab Followed by HCT)
Number analyzed (Participants) | 52
Participants | 14

8. Secondary Outcome: Rituxan Concentration
Description: Median rituxan level at days 60, 84, 180, and 1 year.
Time Frame: Days 60, 84, 180, and 1 year
Population: Number of participants varies by interval based on the number of samples received.14 subjects were enrolled prior to the addition of rituximab. These subjects are counted towards accrual but not evaluated with respect to outcome measures.
Measure: Median (Full Range); unit: ug/ml
Arm/Group | Treatment (Chemotherapy and Rituximab Followed by HCT)
Number analyzed (Participants) | 52
ug/ml
  Day 60: number analyzed (Participants) | 27
  Day 60 | 109 [0.2 to 480.5]
  Day 84: number analyzed (Participants) | 28
  Day 84 | 51 [0.1 to 369]
  Day 180: number analyzed (Participants) | 15
  Day 180 | 1.3 [0 to 103.6]
  1 year: number analyzed (Participants) | 6
  1 year | .03 [0 to 0.6]

9. Secondary Outcome: Number of Patients Achieving Complete Response and Partial Response (Overall Response Rate)
Description: Complete Remission (CR):
  Imaging studies (Xray, CT, MRI) (nodes, liver, and spleen): Normal Peripheral blood by flow cytometry: No clonal lymphocytes Bone marrow by morphology: No nodules; or if present, nodules are free from CLL cells by immunohistochemistry Duration: ≥2 months
  CR with minimal residual disease Peripheral blood or bone marrow by flow cytometry: >0 - <1 CLL cells/1000 leukocytes (0.1%)
  Partial Remission (PR):
  Both criteria:
  Absolute lymphocyte count in peripheral blood: ≥50% decrease Physical exam/Imaging studies (nodes, liver, and/or spleen): ≥50% decrease Duration: ≥2 months
Time Frame: Up to 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy and Rituximab Followed by HCT)
Number analyzed (Participants) | 52
Participants | 35

10. Secondary Outcome: Donor and Host Polymorphisms of the FCgammaRIIIa Receptor and CD32 and Their Impact on Disease Response and Relapse
Description: Number of participants without progressive disease and surviving at one year. Participants with FCgammaRIIIa receptor vs participants without FCgammaRIIIa receptor.
Time Frame: 1 Year
Population: Number of patients with PK sample testing. 14 subjects were enrolled prior to the addition of rituximab. These subjects are counted towards accrual but not evaluated with respect to outcome measures.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy and Rituximab Followed by HCT)
Number analyzed (Participants) | 32
Participants
  Surviving participants w/ FCgammaRIIIa receptor: number analyzed (Participants) | 2
  Surviving participants w/ FCgammaRIIIa receptor | 2
  Surviving participants w/o FCgammaRIIIa receptor: number analyzed (Participants) | 30
  Surviving participants w/o FCgammaRIIIa receptor | 21
  w/ FCgammaRIIIa receptor w/o progressive disease: number analyzed (Participants) | 2
  w/ FCgammaRIIIa receptor w/o progressive disease | 2
  w/o FCgammaRIIIa receptor w/o progressive disease: number analyzed (Participants) | 30
  w/o FCgammaRIIIa receptor w/o progressive disease | 19

ADVERSE EVENTS:
Time Frame: AEs: Conditioning through Day 100; SAEs: Conditioning through Day 200
Description: Historical controls were utilized for comparison
Groups:
- Treatment: Patients receive a conditioning regimen comprising fludarabine IV on days -4 to -2 and rituximab IV on days -3, 10, 24, and 38.
  Patients undergo single fraction low-dose TBI on day 0. After completion of TBI, patients undergo allogeneic hematopoietic stem cell transplantation on day 0. Patients then receive rituximab IV on days 10, 24, and 38.
  Patients receive an immunosuppressive regimen comprising cyclosporine PO BID on days -3 to 56 followed by a taper to day 180 (related recipients) or on days -3 to 100 followed by a taper to day 180 (unrelated recipients). Patients also receive mycophenolate mofetil PO BID on days 0-27 (related recipients) or TID on days 0-40 followed by a taper to day 96 (unrelated recipients).
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo HSCT
  Cyclosporine: Given PO
  Fludarabine Phosphate: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given PO
  Peripheral Blood Stem Cell Transplantation:
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 33/52
Serious Adverse Events (participants affected / at risk) | 4/52
Other Adverse Events (participants affected / at risk) | 22/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=52)
Thrombotic microangiopathy, secondary to cyclosporine, resulting in renal failure requiring dialysis (Renal and urinary disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Death related to grade 4 GVHD (Immune system disorders) | 1 (1)
Death-septic shock related to acute GVHD (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=52)
Volume overload likely precipitating hypoxia and heart failure (Cardiac disorders) | 1 (1)
Chest CT show filling defect that consistent with pulmonary embolism (Cardiac disorders) | 1 (1)
Syncopal episode with neurological exam and head CT unremarkable (Cardiac disorders) | 1 (1)
Decrease in LVEF from 55% to 24% due to volume overload (Cardiac disorders) | 1 (1)
Sharp left sided chest pain (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (3)
Hypotension (Cardiac disorders) | 1 (1)
Weight gain associated with pleural effusion (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Increased bilirubin (Investigations) | 7 (7)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 (7)
Infection (Bacterial & Fungal) (Infections and infestations) | 1 (1)
Syncopal episode (Nervous system disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Creatinine increased (Investigations) | 1 (1)
Systemic inflammatory response syndrome (SIRS) (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-01-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT00104858/Prot_SAP_000.pdf
  • Informed Consent Form (2014-12-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT00104858/ICF_001.pdf